CLINICAL TRIAL: NCT05953532
Title: Developing a Diabetes Self-management mHealth Simulation Platform for Youth
Brief Title: Developing a mHealth Simulation Platform for Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022N0018
Record Dates: First submitted 2023-06-13; First posted 2023-07-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Engagement, Patient
MeSH Terms: conditions — Patient Participation

STUDY DESIGN:
Intervention Model Description: Single group pilot study to evaluate youth engagement
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All Participants (Other): All participants will perform the same study activities
  Interventions: Other: A1Control

INTERVENTIONS:
Other: A1Control — diabetes self-management and diabetes technology education software

SUMMARY:
The investigators will conduct a 12-week single group feasibility pilot field study among youth who will use a diabetes technology education application in their natural home environment.

DETAILED DESCRIPTION:
The investigators will purposively select N=20 youth with at least 6 youth from each of 3 age ranges (10-12, 13-15, and 16-18) from eligible participants. Youth will use the software in their home environment for 12-weeks. Youth's diabetes device data will be used to select simulation content, targeted to meet each participant's educational needs. Youth will meet with research staff via video chat at the onset of testing where a URL link to the platform will be shared. Youth will be assigned 3 scenarios/week. At the end of each scenario youth are guided to additional resources in the platform that they may choose to access. Youth will meet with a member of the research team via video chat or phone call weekly to discuss platform issues or confusion as well as any questions regarding self-management content. Platform performance will be monitored by researchers and performance data will be collected and stored within the application database.

Feasibility measures will include recruitment, weekly research sessions attendance, and global attrition data. Sustained engagement measures will be collected from the application database and will include the frequency platform was accessed, number of assigned simulations completed (3 per week), and additional, optional, content accessed. Glycemic control measures including A1C will be obtained from the youth's EHR. Youth's diabetes devices will be downloaded at baseline and at 4, 6 and 12 weeks. Glucose values from device downloads will be aggregated into derived measures of glucose control consistent with American Diabetes Association guidelines on glucose targets. Self-management patterns and responsiveness will be assessed using pre- and post- diabetes device downloads at baseline, 4, 8, and 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 1 diabetes >1 year
* 10-18 years of age
* Currently uses insulin pump or HCL therapy
* Duration of 6 months of pump therapy

Exclusion Criteria:

* Significant learning disability
* Self-reported pregnancy
* Inability to read and write English

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Measure of Engagement in Personal Healthcare | 12-weeks
  frequency that the platform is accessed by the participant, number of assigned simulations scenarios completed (out of 3 assigned per week), and additional, optional, content accessed by the participant

SECONDARY OUTCOMES:
Glycemic control | baseline, 4, 8, and 12 weeks
  Percent time spent in target glucose range (70-180mg/dl)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Nationwide Children's Hospital, Columbus, Ohio
  - The Ohio State University, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No